CLINICAL TRIAL: NCT06432842
Title: Knee Osteoarthritis and Lazer Therapy
Brief Title: Knee Osteoarthritis and Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, METEHAN YANA, Director, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Karabuk-80
Record Dates: First submitted 2024-03-25; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Knee Osteoarthritis
Keywords: Osteoarthritis; Intra-articular injection; PRP (Platelet-rich plasma); Physiotherapy; Laser Treatment
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Laser Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional treatment (Active Comparator): Within the scope of conventional treatment, individuals were given Transcutaneous Electrical Nerve Stimulation (TENS), infrared, US and exercise therapy.
  Interventions: Other: Laser Treatment
- Laser treatment (Active Comparator): In the study group, low-dose laser treatment was applied in addition to conventional treatment. Therapeutic Laser device was used for laser treatment. Laser treatment was applied to 8 sensitive points around the knee for 1 minute, for a total of 8 minutes.
  Interventions: Other: Laser Treatment

INTERVENTIONS:
Other: Laser Treatment — In the study group, low-dose laser treatment was applied in addition to conventional treatment. Chattanoga Group Therapeutic Laser device was used for laser treatment. Laser treatment was applied to 8 sensitive points around the knee for 1 minute, for a total of 8 minutes. Laser treatment was applied continuously, with a wavelength of 830nm and a power of 6J.
  Other Names: conventional treatment

SUMMARY:
Osteoarthritis (OA) is a chronic degenerative disease of articular cartilage that causes hypertrophic changes in bone. OA is a non-inflammatory progressive musculoskeletal disease and is one of the most common degenerative diseases in the general population. OA is characterized by progressive cartilage destruction in load-bearing joints, subchondral sclerosis, osteophyte formation, and some biochemical and morphological changes in the synovial membrane and joint capsule. Common symptoms of knee osteoarthritis are; Knee pain that increases with activity, limitation of normal joint movement of the knee, edema, and knee pain that begins with prolonged sitting.

The aim of this study is to evaluate the effects of laser treatment applied in addition to conventional physiotherapy on pain, function, muscle strength and balance in patients with knee osteoarthritis who received PRP.

DETAILED DESCRIPTION:
OA is a non-inflammatory progressive musculoskeletal disease; damage begins in the cartilage and causes changes in the joint structure over time. Although intra-articular injection approaches have been frequently used in the treatment of OA recently, intra-articular injections known as Platelet Rich Plasma (PRP) have also started to be used frequently. Today, the areas of use of laser therapy have increased. When the laser beam is applied, it is absorbed by the tissue or scattered back. Laser has photochemical, thermal and ionizing effects on tissues. Laser has an analgesic effect by increasing endorphin synthesis and reducing C nerve fiber activation. Laser indirectly increases microcirculation by increasing temperature in the tissue. Although there are various studies on treatment options for OA in the literature, no studies have been found to investigate the effectiveness of laser treatment applied in addition to conventional treatment after PRP. In our study, we aimed to evaluate the effects of laser treatment applied in addition to conventional physiotherapy on pain, function, muscle strength and balance in patients with knee osteoarthritis who received PRP.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Being diagnosed with knee OA by a specialist physician
* Having had PRP injection applied by a specialist physician
* Having unilateral knee OA
* Being stage I-stage III in the Kellgren-Lawrence OA classification
* Being between the ages of 18-65

Exclusion Criteria:

* Being stage IV in the Kellgren-Lawrence OA classification
* BMI being more than 40 kg/m2
* Patients who do not cooperate well
* Patients with neurological or neuromuscular disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain severity | Baseline and 2 weeks post-intervention
  Knee pain severity will measured using the Visual Analog Scale. Scale (VAS). The VAS is a 10 cm scale, where 0 represented no pain and 10 represented unbearable pain. Pain intensity was recorded by measuring the point marked between 0- 10.
Function | 2 weeks post-intervention
  WOMAC will be used to evaluate the degree of physical function. This scale has a total of 24 questions and 5 answers between 0-4 for each question. A high score indicates that the symptoms are severe.
MUSCLE STRENGTH | Baseline and 2 weeks post-intervention
  Hip, knee flexor and extensor muscle strengths will be measured using a manual dynamometer.
BALANCE | Baseline and 2 weeks post-intervention
  Dynamic balance of individuals through the Modified Star Balance Test will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Karabük University, Karabük, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fitzgerald GK, Piva SR, Irrgang JJ. Reports of joint instability in knee osteoarthritis: its prevalence and relationship to physical function. Arthritis Rheum. 2004 Dec 15;51(6):941-6. doi: 10.1002/art.20825. PMID 15593258
- [Background] Fransen M, McConnell S, Harmer AR, Van der Esch M, Simic M, Bennell KL. Exercise for osteoarthritis of the knee: a Cochrane systematic review. Br J Sports Med. 2015 Dec;49(24):1554-7. doi: 10.1136/bjsports-2015-095424. Epub 2015 Sep 24. PMID 26405113
- [Background] Hedbom E, Hauselmann HJ. Molecular aspects of pathogenesis in osteoarthritis: the role of inflammation. Cell Mol Life Sci. 2002 Jan;59(1):45-53. doi: 10.1007/s00018-002-8404-z. PMID 11846032
- [Background] Citaker S, Gunduz AG, Guclu MB, Nazliel B, Irkec C, Kaya D. Relationship between foot sensation and standing balance in patients with multiple sclerosis. Gait Posture. 2011 Jun;34(2):275-8. doi: 10.1016/j.gaitpost.2011.05.015. Epub 2011 Jun 16. PMID 21683600
- [Background] Chapple CM, Nicholson H, Baxter GD, Abbott JH. Patient characteristics that predict progression of knee osteoarthritis: a systematic review of prognostic studies. Arthritis Care Res (Hoboken). 2011 Aug;63(8):1115-25. doi: 10.1002/acr.20492. PMID 21560257
- [Background] MILLER JH, WHITE J, NORTON TH. The value of intra-articular injections in osteoarthritis of the knee. J Bone Joint Surg Br. 1958 Nov;40-B(4):636-43. doi: 10.1302/0301-620X.40B4.636. No abstract available. PMID 13610976
- [Background] McAlindon TE, Bannuru RR, Sullivan MC, Arden NK, Berenbaum F, Bierma-Zeinstra SM, Hawker GA, Henrotin Y, Hunter DJ, Kawaguchi H, Kwoh K, Lohmander S, Rannou F, Roos EM, Underwood M. OARSI guidelines for the non-surgical management of knee osteoarthritis. Osteoarthritis Cartilage. 2014 Mar;22(3):363-88. doi: 10.1016/j.joca.2014.01.003. Epub 2014 Jan 24. PMID 24462672
- [Background] Hagiwara S, Iwasaka H, Okuda K, Noguchi T. GaAlAs (830 nm) low-level laser enhances peripheral endogenous opioid analgesia in rats. Lasers Surg Med. 2007 Dec;39(10):797-802. doi: 10.1002/lsm.20583. PMID 18081143
- [Background] Raeissadat SA, Rayegani SM, Hassanabadi H, Fathi M, Ghorbani E, Babaee M, Azma K. Knee Osteoarthritis Injection Choices: Platelet- Rich Plasma (PRP) Versus Hyaluronic Acid (A one-year randomized clinical trial). Clin Med Insights Arthritis Musculoskelet Disord. 2015 Jan 7;8:1-8. doi: 10.4137/CMAMD.S17894. eCollection 2015. PMID 25624776